CLINICAL TRIAL: NCT02026466
Title: Outcomes, Patient Health Status, and Efficiency in Chronic Total Occlusion (OPEN CTO)
Brief Title: Outcomes, Patient Health Status, and Efficiency in Chronic Total Occlusion
Acronym: OPEN-CTO
Status: Completed | Type: Observational
Sponsor: Saint Luke's Health System (Other)
Collaborators: Boston Scientific Corporation (Industry)
Responsible Party: Sponsor
Other Study IDs: OPEN CTO V1.2
Record Dates: First submitted 2013-11-26; First posted 2014-01-03 (Estimated); Last update posted 2021-10-19 (Actual); Status verified 2021-10

CONDITIONS: Coronary Artery Disease
Keywords: Coronary Artery Disease; Chronic Total Occlusion
MeSH Terms: conditions — Coronary Artery Disease

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 5 Years
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- CAD with CTO: Subjects will have Coronary Artery Disease with a diagnosed Chronic Total Occlusion: a coronary artery with TIMI flow of zero(no flow) for at least three months.

SUMMARY:
This is an observational registry, sponsored by Saint Luke's Hospital. This study is to be conducted according to DHHS Guidelines, applicable state regulations, and local IRB policies and procedures. The overall objective is to address current gaps in knowledge regarding CTO-PCI, as a prospective, multi-center, single-arm study of 1,000 participants.

DETAILED DESCRIPTION:
* 1,000 participants will be enrolled into the OPEN CTO study.
* Study coordinators will screen both men and women over the age of 18 who are admitted for an elective CTO-PCI procedure.
* Study coordinators will be trained by the Coordinating Center at Saint Luke's Hospital of Kansas City.
* Participants will be screened for Eligibility, and Informed Consent will be obtained.
* Participants will also be asked to sign a Medical Records Release form, and a Billing Records Release form.
* Detailed procedural data will be obtained by the Study Coordinator and local Principal Investigator.
* Participants will undergo a Baseline interview.
* These data will be entered into the electronic data capture system, Velos, which has stringent protections and quality controls.
* Participants will have telephone follow-up interviews conducted by the centralized Follow-up Center at Saint Luke's Hospital.

ELIGIBILITY:
Inclusion Criteria:

* Subject is scheduled for a PCI procedure for at least one chronic total occlusion with TIMI antegrade flow of zero.
* Subject is ≥ 18 years of age at the time of consent.

Exclusion Criteria:

* The CTO segment is in a graft
* Female subjects with a positive quantitative or qualitative pregnancy test, in accordance with hospital policy.
* Non-English speaking
* Too hard of hearing to do follow-up by telephone.
* Previously enrolled in OPEN CTO Registry
* Currently a prisoner
* Dementia
* Subjects with no way contact by telephone for follow-up.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: 18 or older with CAD and at least one chronic total occluded vessel.
Sampling Method: Non-Probability Sample
Enrollment: 1000 (Actual)
Dates: Start 2013-12 (Actual); Primary Completion 2017-09 (Actual); Study Completion 2017-12 (Actual)

PRIMARY OUTCOMES:
Health Status | One year
  Quantify the baseline health status effects of CTO among patients selected for CTO-PCI and quantify the changes associated with CTO-PCI using the Hybrid Approach.

SECONDARY OUTCOMES:
Safety and Effectiveness | One Year
  Describe safety and effectiveness among patients receiving CTO-PCI

CONTACTS AND LOCATIONS:
Overall Officials: J. Aaron Grantham, MD, Principal Investigator — Saint Luke's Health System
Locations (11):
- United States (11):
  - Banner Heart Hospital, Mesa, Arizona
  - Banner Good Samaritan, Phoenix, Arizona
  - Torrance Memorial Medical Center, Torrance, California
  - Alexian Brothers Medical Center, Elk Grove Village, Illinois
  - Boone Hospital Center, Columbia, Missouri
  - Saint Luke's Hospital of Kansas City, Kansas City, Missouri
  - Presbyterian Health System Hospital, Albuquerque, New Mexico
  - Columbia University Medical Center, New York, New York
  - Peace Health Sacred Heart River Bend Medical Center, Springfield, Oregon
  - York Hospital, York, Pennsylvania
  - University of Washington Medical Center, Seattle, Washington

REFERENCES:
- [Result] Brilakis ES, Grantham JA, Rinfret S, Wyman RM, Burke MN, Karmpaliotis D, Lembo N, Pershad A, Kandzari DE, Buller CE, DeMartini T, Lombardi WL, Thompson CA. A percutaneous treatment algorithm for crossing coronary chronic total occlusions. JACC Cardiovasc Interv. 2012 Apr;5(4):367-79. doi: 10.1016/j.jcin.2012.02.006. PMID 22516392
- [Derived] Hirai T, Qintar M, Grantham JA, Sapontis J, Cohen DJ, Lombardi W, Karmpaliotis D, Moses J, Nicholson WJ, Nugent K, Gosch KL, Spertus JA, Salisbury AC. Patient Characteristics Associated With Antianginal Medication Escalation and De-Escalation Following Chronic Total Occlusion Percutaneous Coronary Intervention. Circ Cardiovasc Qual Outcomes. 2019 Jun;12(6):e005287. doi: 10.1161/CIRCOUTCOMES.118.005287. Epub 2019 Jun 12. PMID 31185735
- [Derived] Yeh RW, Tamez H, Secemsky EA, Grantham JA, Sapontis J, Spertus JA, Cohen DJ, Nicholson WJ, Gosch K, Jones PG, Valsdottir LR, Bruckel J, Lombardi WL, Jaffer FA. Depression and Angina Among Patients Undergoing Chronic Total Occlusion Percutaneous Coronary Intervention: The OPEN-CTO Registry. JACC Cardiovasc Interv. 2019 Apr 8;12(7):651-658. doi: 10.1016/j.jcin.2018.12.029. Epub 2019 Mar 13. PMID 30878475